CLINICAL TRIAL: NCT06578858
Title: Immunonutrition and Psychosocial Factors in the Recovery of Patients After Gastric Cancer Surgery: a Multidimensional Analysis
Brief Title: Immunonutrition and Psychosocial Factors in the Recovery of Patients After Gastrectomy: a Multidimensional Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Igor Gabriel Araújo Medeiros, Student at the Federal University of Pernambuco, Universidade Federal de Pernambuco
Other Study IDs: 81097524.9.0000.5208
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Salutogenesis; Sense of Coherence
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Application of questionnaires — Application of SOC-13 and BRS questionnaires in patients after gastric cancer surgery

SUMMARY:
To conduct this research, the following guiding question was formulated: "Can immunonutrition, combined with the assessment of SOC and resilience, provide a broad view of the physical and psychological results during the treatment and recovery process of patients undergoing gastric cancer surgery?". This led to the formulation of the following hypothesis: "Patients who received immunonutrition and who have higher levels of resilience and sense of coherence will tend to exhibit more favorable clinical and laboratory outcomes for recovery after gastric cancer surgery.

In order to answer the question and test the study hypothesis, the general objective consisted of:

To evaluate the association of clinical and laboratory outcomes with the sense of coherence and resilience of patients undergoing gastric cancer surgery who received immunonutrition.

In view of this general objective, the following specific objectives were formulated:

* To evaluate the levels of resilience and sense of coherence in patients undergoing gastric cancer surgery who received immunonutrition.
* Analyze the results of blood count and C-Reactive Protein (CRP) in patients who received immunonutrition after gastric cancer surgery.
* Identify the association between resilience levels, sense of coherence, blood count and CRP values with clinical outcomes, such as length of hospital stay and wound recovery, in patients undergoing gastric cancer surgery who used immunonutrition.

ELIGIBILITY:
Inclusion Criteria:

Adult or elderly patients (age ≥ 18 years) Treated at Consultório Guararapes Underwent surgery to remove gastric cancer Used immunonutrition in the pre, post, or perioperative period Applicable to both sexes

Exclusion Criteria:

Pre-existing hematologic diseases that may affect blood count results History of drug abuse (legal and/or illegal) Presence of other neoplasms History of psychological disorders affecting ability to respond to study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have undergone gastric cancer removal surgery and used immunonutrition in the pre or perioperative period
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Resilience Levels and Clinical Outcomes | Questionnaires to assess resilience and sense of coherence will be administered once, after gastric cancer removal surgery.
  1) Separate outcome measures:
  Levels of resilience Title: Measure of resilience level Description: Resilience will be measured using the Resilience Scale, with scores ranging from (1.00 - 2.99) = Low; (3.00 - 4.30) = Normal; (4.31 - 5.00) = High Unit of measurement: Score Measurement tool: Brief Resilience Scale (BRS)
  Sense of coherence Title: Measure of sense of coherence Description: Sense of coherence will be assessed using the Sense of coherence Scale, with a median of 35 Unit of measurement: Median (35) Measurement tool: Sense of coherence scale questionnaire (SOC-13)

CONTACTS AND LOCATIONS:
Locations (1):
- Consultorios Guararapes, Jaboatão dos Guararapes, Pernambuco, Brazil